CLINICAL TRIAL: NCT07325071
Title: A Randomized Controlled Trial Comparing Conventional and Short Submucosal Tunnel Techniques in Type II Achalasia
Brief Title: Comparison of Conventional and Short Submucosal Tunnel Techniques in Type II Achalasia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, MD, DM, FJGES , Director interventional Endoscopy , senior consultant Gastroenterologist, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRIM POEM
Record Dates: First submitted 2025-09-27; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Esophageal Diseases
MeSH Terms: conditions — Esophageal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Control Group) (Other): Conventional POEM with 10-12 cm submucosal tunnel, 6-8 cm Esophageal myotomy, and 2 cm gastric myotomy
  Interventions: Procedure: Arm A - Conventional POEM (Control Arm)
- Arm B (Standard Submucosal Tunnel + EGJ - complex only Myotomy) (Active Comparator): 10-12 cm submucosal tunnel with myotomy restricted to the EGJ (2 cm Esophageal and 2 cm gastric)
  Interventions: Procedure: Arm B - Standard Tunnel with EGJ complex-only Myotomy; Procedure: Arm C - Ultra-short Tunnel POEM with EGJ complex -only Myotomy
- Arm C (Ultra-short Tunnel + EGJ- complex only Myotomy) (Active Comparator): 4 cm submucosal tunnel with myotomy focused on the EGJ (2 cm Esophageal and 2 cm gastric)
  Interventions: Procedure: Arm B - Standard Tunnel with EGJ complex-only Myotomy; Procedure: Arm C - Ultra-short Tunnel POEM with EGJ complex -only Myotomy

INTERVENTIONS:
Procedure: Arm A - Conventional POEM (Control Arm) — Arm A - Conventional POEM (Control Arm)
  * Tunnel Length: 10-12 cm submucosal tunnel, extending from 10 cm proximal to the EGJ into the proximal stomach.
  * Myotomy:
    * Esophageal segment: 6-8 cm
    * Gastric segment: 2 cm
    * Myotomy orientation: posterior (5-6 o'clock position)
    * Depth: selective circular myotomy in Esophageal segment, full-thickness at LES and gastric side
  Arms: Arm A (Control Group)
Procedure: Arm B - Standard Tunnel with EGJ complex-only Myotomy — * Tunnel Length: 10-12 cm submucosal tunnel to allow full-length inspection and safe scope manipulation.
  * Myotomy:
    * Esophageal: 2 cm proximal to EGJ
    * Gastric: 2 cm distal to EGJ
    * Purpose: limit disruption of Esophageal muscle above EGJ while retaining effective LES division
    * Myotomy is confined to the EGJ complex while still using a standard tunnel
    * Full-thickness myotomy may be used at the EGJ for consistency
  Arms: Arm B (Standard Submucosal Tunnel + EGJ - complex only Myotomy); Arm C (Ultra-short Tunnel + EGJ- complex only Myotomy)
Procedure: Arm C - Ultra-short Tunnel POEM with EGJ complex -only Myotomy — * Tunnel Length: Approximately 4 cm, just enough to reach the EGJ complex and enable targeted dissection
  * Myotomy:
    * Esophageal: 2 cm
    * Gastric: 2 cm
    * Only the EGJ segment is divided, minimising disruption of proximal Esophageal musculature
    * Myotomy is performed selectively along the posterior axis (5-6 o'clock) Intraoperative Assessment and Quality Control
  * Adequacy of gastric extension is confirmed with visualisation of retroflexed scope or via second scope trans illumination when needed.
  * Any bleeding is controlled with coagulation graspers or cautery.
  * Tunnelling is performed closely along the Muscularis propria to minimise mucosal injury.
  * The scope is periodically withdrawn for mucosal inspection during the procedure.
  Arms: Arm B (Standard Submucosal Tunnel + EGJ - complex only Myotomy); Arm C (Ultra-short Tunnel + EGJ- complex only Myotomy)

SUMMARY:
Rationale for This Study The primary rationale for this study is to evaluate whether a shorter submucosal tunnel during POEM with an EGJ-focused myotomy in type II Achalasia cardia patients, provides equivalent or superior symptom relief compared to the conventional approach while minimizing adverse events such as GERD & blown out myotomy and decreasing the procedure time.

Objectives

Primary Objective:

To compare the incidence of GERD (with manual review) at 3 and 12 months' post-procedure between conventional POEM and two experimental short-tunnel POEM techniques in patients with Type II achalasia.

Secondary Objectives:

To evaluate

1. Clinical success based on Eckardt score
2. Operating total procedure time
3. Use of Acid Suppressants on Follow up at 1 year
4. Severity of Esophagitis at 3 months
5. Intraoperative & Postoperative adverse events (AGREE classification),
6. GERD-HRQL (0-18) scores 3 & 12 Months
7. (Clinically relevant GORD was defined as excessive oesophageal /AET associated with a GERDQ score >7 and/or with any grade of reflux oesophagitis).
8. Duration of Hospital stay
9. Quality of life (SF36)

DETAILED DESCRIPTION:
Achalasia type II is the most common manometric subtype and responds well to Peroral Endoscopic Myotomy (POEM). However, the optimal extent of submucosal tunneling and myotomy length for this population remains uncertain. Conventional POEM typically involves a 10-12 cm submucosal tunnel with a long esophageal myotomy (6-8 cm) and a 2-3 cm gastric extension. While effective, this approach may predispose patients to higher rates of post-procedure gastroesophageal reflux disease (GERD), mucosal injuries, and CO₂-related insufflation events due to more extensive dissection.

Recent physiologic data from FLIP studies suggest that disrupting the esophagogastric junction (EGJ) complex alone-approximately 2 cm proximally and 2-3 cm distally-may be sufficient to normalize EGJ distensibility in achalasia. Additional proximal myotomy does not appear to improve compliance and may unnecessarily increase the risk of adverse events or compromise esophageal motor recovery. Emerging randomized studies have further shown that shorter esophageal myotomies (≤5 cm) can provide symptom relief comparable to standard approaches, with potentially lower reflux rates.

This trial evaluates whether limiting myotomy to the EGJ complex, with or without a shorter submucosal tunnel, can reduce post-POEM GERD while maintaining clinical efficacy in Type II achalasia. The study uses a three-arm randomized controlled design comparing:

Conventional POEM with long submucosal tunnel and long esophageal myotomy;

Standard-length tunnel with EGJ-only myotomy, preserving proximal esophageal muscle while maintaining full tunnel access;

Ultra-short tunnel POEM with EGJ-only myotomy, minimising dissection length and procedure time.

All procedures follow standardized POEM steps, including mucosal entry, submucosal tunneling, myotomy, and mucosal closure. Technical variations between arms are restricted to tunnel length and myotomy extent. Myotomy is performed primarily on the posterior axis, with selective circular myotomy proximally and full-thickness division across the LES as clinically appropriate. Adequacy of gastric extension is confirmed visually, and all mucosal incisions are closed using through-the-scope clips. Intraoperative quality control measures include frequent mucosal inspection, careful dissection along the muscularis propria, and standard management of bleeding or capnoperitoneum.

Participants are randomized in a 1:1:1 ratio using concealed allocation. Blinding of operators is not feasible, but outcome assessors, data collectors, and statisticians remain blinded to minimize detection and assessment bias. Post-procedure evaluation includes symptomatic scoring, endoscopy, manometry when applicable, and 24-hour pH impedance testing. GERD will be assessed both physiologically and via validated patient-reported measures. Adverse events will be systematically recorded using the AGREE classification.

An independent Data and Safety Monitoring Board will conduct an interim analysis after 50% of participants complete 3-month follow-up, with pre-specified stopping rules for superiority, futility, or harm. The large sample size and three-arm design are intended to allow detection of clinically meaningful differences in GERD incidence while ensuring the trial remains adequately powered after accounting for anticipated non-compliance.

This study aims to provide high-quality, comparative data on whether submucosal tunnel length and targeted myotomy at the EGJ can optimize outcomes for Type II achalasia. If shorter techniques demonstrate equivalent clinical success with lower GERD rates and fewer adverse events, they may represent a safer and more efficient modification of the standard POEM procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged >18 years.
2. Diagnosis of Type II achalasia naïve patients based on high-resolution manometry (Chicago Classification v4).
3. Eckardt score >3.
4. Written informed consent

Exclusion Criteria:

1. Type I or III achalasia.
2. Previous endoscopic or surgical treatment for achalasia.
3. Contraindications for POEM (e.g., coagulopathy, portal hypertension).
4. Sigmoid Achalasia

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-06-20 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Gastro esophageal Reflux disease (GERD) after poem | At 12 weeks and 52 weeks post-procedure
  Comparison of gastroesophageal reflux disease incidence, assessed by manual review of esophageal acid exopsure and endoscopic findings, between conventional poem and two experimental short tunnel poem techinques in patients with type II achalasia

SECONDARY OUTCOMES:
Eckardt symptom score | At 12 weeks and 52 weeks post-procedure
  Clinical success assessed using the Eckardt Symptom Score, a validated symptom scoring system for achalasia.
  Scale range: 0 to 12
  Score < 3 indicates clinical success
  Higher scores indicate worse symptoms
Total procedure time | Periprocedural (during the procedure)
  Total duration of the POEM procedure measured from mucosal incision to mucosal closure, recorded in minutes.
use of acid suppressants | Up to 1 year post-procedure
  Requirement for acid suppressive medications, including proton pump inhibitors (PPIs) or H2-receptor blockers, following the procedure.
severity of esophagitis | At 12 weeks post procedure
  Severity of esophagitis assessed by upper gastrointestinal endoscopy using the Los Angeles Classification of Esophagitis:
  Scale:
  Grade A = mild Grade B = moderate Grade C = severe Grade D = very severe (Higher grades indicate more severe esophagitis.)
intraoperative and post operative adverse events | Periprocedural and post-procedure
  Intraoperative and postoperative complications classified according to the AGREE Classification, graded from A to E, where higher grades indicate more severe adverse events.Grades A to E Higher grades indicates more adverse events
Gastroesophageal Reflux Disease- Health Related Quality of Life questionnaire (GERD-HRQL) | At 12 weeks and 52 weeks post-procedure
  Patient-reported gastroesophageal reflux disease-related quality of life assessed using the Gastroesophageal Reflux Disease- Health Related Quality of Life questionnaire.
  Scale range: 0 to 18
  Higher scores indicate worse Gastroesophageal Reflux Disease-related quality of life
Clinically relevant Gastroesophageal Reflux Disease Questionnaire (GERD-Q) | At 1 year post-procedure
  Clinically relevant GERD assessed using the Gastroesophageal Reflux Disease Questionnaire (GERD-Q).
  Scale range: 0 to 18 Higher scores indicate worse Gastroesophageal Reflux Disease symptoms Clinically relevant Gastroesophageal Reflux Disease defined as Gastroesophageal Reflux Disease Questionnaire (GERD-Q). score > 7 and/or presence of reflux esophagitis on endoscopy with abnormal esophageal acid exposure time (AET)
duration of hospital stay | up to 1 week
  Length of hospital stay measured as the total number of inpatient days following the procedure.
36-Item Short Form Survey (SF-36) | At baseline (pre-procedure), 12 weeks, and 52 weeks post-procedure
  Health-related quality of life assessed using the 36-Item Short Form Health Survey (SF-36).
  Scores range from 0 to 100 for each domain Higher scores indicate better health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Mohan Kumar Ramchandani, MD, DM, Study Director — AIG Hospitals

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nabi Z, Talukdar R, Mandavdhare H, Reddy DN. Short versus long esophageal myotomy during peroral endoscopic myotomy: A systematic review and meta-analysis of comparative trials. Saudi J Gastroenterol. 2022 Jul-Aug;28(4):261-267. doi: 10.4103/sjg.sjg_438_21. PMID 34806659
- [Result] Stefanidis D, Richardson W, Farrell TM, Kohn GP, Augenstein V, Fanelli RD; Society of American Gastrointestinal and Endoscopic Surgeons. SAGES guidelines for the surgical treatment of esophageal achalasia. Surg Endosc. 2012 Feb;26(2):296-311. doi: 10.1007/s00464-011-2017-2. Epub 2011 Nov 2. No abstract available. PMID 22044977